CLINICAL TRIAL: NCT00492544
Title: Evaluation of the Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV Vaccine 580299 When Administered as a 3-dose Schedule in Healthy Japanese Pre-adolescent and Adolescent Female Subjects.
Brief Title: Immunogenicity and Safety of GSK Biologicals' HPV Vaccine 580299 in Healthy Japanese Females 10-15 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 110168
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2009-12-21 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Infections, Papillomavirus
Keywords: Human Papillomavirus (HPV) vaccine; safety; cervical cancer; immunogenicity; vaccine; viral infections; pre-adolescent and adolescent females
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Virus Diseases | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- Cervarix (Experimental): Subjects received 3 doses of Cervarix™ (HPV-16/18 L1 VLP AS04) according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix™ (HPV-16/18 L1 VLP AS04)

INTERVENTIONS:
Biological: Cervarix™ (HPV-16/18 L1 VLP AS04) — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Other Names: GSK Biologicals' HPV-16/18 VLP/AS04 vaccine

SUMMARY:
Human papillomavirus (HPV) infection has been established as a necessary cause of cervical cancer. GSK Biologicals has developed an HPV vaccine (580299) which targets the 2 most common oncogenic HPV types (HPV-16 and HPV-18), found in approximately 70% of all cervical cancers. In previous trials, the vaccine has been found to be efficacious in the prevention of incident and persistent HPV-16/18 infections and associated cytological abnormalities. HPV vaccination should ideally be performed before onset of sexual activity. Previous studies showed that GSK Biologicals' HPV vaccine 580299 is safe and immunogenic when administered to European, Asian, Latin American and Australian pre-adolescents and adolescents. Here, we aim to assess the immunogenicity and safety of the GSK Biologicals' HPV vaccine 580299 in healthy Japanese pre-adolescent and adolescent female subjects aged 10-15 years. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator/co-investigator believes that they and/or their parent(s)/legally acceptable representative(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* A Japanese female between, and including, 10 and 15 years of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s) or legally acceptable representative(s) of the subject. In addition, a written informed assent must be obtained from the subject prior to enrolment.
* Healthy subjects as established by medical history and history-directed clinical examination before entering into the study.
* All subjects must have a negative urine pregnancy test.
* Subjects must be of non-childbearing potential, or, if of childbearing potential, they must be abstinent or have used adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series. Non-abstinent pre-menarche subjects, as well as subjects who reach menarche during study, must follow the same precautions.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned during study.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. Administration of vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period (up to Month 7), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period (Day 0 to Month 7).
* Previous administration of components of the investigational vaccine .
* Cancer or autoimmune disease under treatment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or breastfeeding subject.
* Subject planning to become pregnant or planning to discontinue contraceptive precautions.
* Oral temperature ≥ 37.5°C/Axillary temperature ≥ 37.5°C.

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-07-02 (Actual); Primary Completion 2008-03-28 (Actual); Study Completion 2008-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Japan (2):
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110168 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervarix Group: Subjects received 3 doses of Cervarix™ (HPV-16/18 L1 VLP AS04) according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the sera of subjects seronegative before vaccination.
  Cut-off values were 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: One month post Dose 3 (Month 7)
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 94
Participants
  Anti-HPV-16: number analyzed (Participants) | 92
  Anti-HPV-16 | 92
  Anti-HPV-18 | 94

2. Primary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) calculated on all subjects.
Time Frame: Before vaccination (PRE) and one month post Dose 3 (Month 7)
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix Group
Number analyzed (Participants) | 99
titer
  Anti-HPV-16 (PRE) | 4.4 [4.1 to 4.8]
  Anti-HPV-16 (Month 7) | 19748.0 [17147.7 to 22742.7]
  Anti-HPV-18 (PRE): number analyzed (Participants) | 98
  Anti-HPV-18 (PRE) | 3.7 [3.5 to 3.9]
  Anti-HPV-18 (Month 7): number analyzed (Participants) | 98
  Anti-HPV-18 (Month 7) | 8765.3 [7543.8 to 10184.4]

3. Primary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 7-day (Days 0-6) period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Participants
  Pain | 98
  Redness | 85
  Swelling | 81

4. Primary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, fever, gastrointestinal symptoms, headache, myalgia, rash, and urticaria.
Time Frame: During the 7-day (Days 0-6) period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Participants
  Arthralgia | 15
  Fatigue | 40
  Fever | 10
  Gastrointestinal symptoms | 17
  Headache | 33
  Myalgia | 26
  Rash | 5
  Urticaria | 3

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: Unsolicited adverse event= Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 30-day (Days 0-29) period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Participants | 63

6. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Other Medically Significant Conditions
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes. Medically significant conditions assessed include adverse events prompting emergency room visits and physician office visits not related to common illnesses or Serious Adverse Events that are not related to common illnesses.
Time Frame: From Day 0 up to Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Participants
  NOCDs | 0
  Medically significant conditions | 18

7. Secondary Outcome: Outcome of All Pregnancies
Description: According to the study protocol, the outcome of all pregnancies reported during the entire study period was to be reported, even if delivery occurs after the end of the study.
Time Frame: Up to Month 7
Population: There were no pregnancies reported between Day 0 and Month 7 in the Total Vaccinated Cohort.
Arm/Group | Cervarix Group
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: Serious adverse events assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Participants | 0

9. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Parameters
Description: Abnormalities include values outside (above or below) the normal ranges.
  Normal ranges:
  alanine aminotransferase (ALT): 5-35 U/L aspartate aminotransferase (AST): 5-50 U/L basophils: 0-2 % bilirubin total: 0.1-1.1 mg/dL blood urea nitrogen: 0-20 mg/dL creatinine: 0.2-1.2 mg/dL eosinophils: 0-7 % hematocrit: 30-45 % hemoglobin: 10-15 g/dL lymphocytes: 18-50 % monocytes: 1-8 % neutrophils: 42-74 % platelets: 10-60 10E4/microL red blood cells: 350-550 10E4/microL total protein: 6.5-8.6 g/dL white blood cells: 4000-15000 /microL
Time Frame: At Day 0 and Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 100
Participants
  ALT Above (Day 0) | 2
  ALT Below (Day 0) | 0
  ALT Above (Month 7) | 1
  ALT Below (Month 7) | 0
  AST Above (Day 0) | 0
  AST Below (Day 0) | 0
  AST Above (Month 7) | 1
  AST Below (Month 7) | 0
  Basophils Above (Day 0) | 0
  Basophils Below (Day 0) | 0
  Basophils Above (Month 7) | 0
  Basophils Below (Month 7) | 0
  Blood urea nitrogen Above (Day 0) | 2
  Blood urea nitrogen Below (Day 0) | 0
  Blood urea nitrogen Above (Month 7) | 0
  Blood urea nitrogen Below (Month 7) | 0
  Creatinine Above (Day 0) | 0
  Creatinine Below (Day 0) | 0
  Creatinine Above (Month 7) | 0
  Creatinine Below (Month 7) | 0
  Eosinophils Above (Day 0) | 17
  Eosinophils Below (Day 0) | 0
  Eosinophils Above (Month 7) | 8
  Eosinophils Below (Month 7) | 0
  Hematocrit Above (Day 0) | 2
  Hematocrit Below (Day 0) | 0
  Hematocrit Above (Month 7) | 0
  Hematocrit Below (Month 7) | 1
  Hemoglobin Above (Day 0) | 0
  Hemoglobin Below (Day 0) | 0
  Hemoglobin Above (Month 7) | 1
  Hemoglobin Below (Month 7) | 1
  Lymphocytes Above (Day 0) | 13
  Lymphocytes Below (Day 0) | 0
  Lymphocytes Above (Month 7) | 4
  Lymphocytes Below (Month 7) | 0
  Monocytes Above (Day 0) | 1
  Monocytes Below (Day 0) | 0
  Monocytes Above (Month 7) | 13
  Monocytes Below (Month 7) | 0
  Neutrophils Above (Day 0) | 0
  Neutrophils Below (Day 0) | 21
  Neutrophils Above (Month 7) | 0
  Neutrophils Below (Month 7) | 7
  Platelets Above (Day 0) | 0
  Platelets Below (Day 0) | 0
  Platelets Above (Month 7) | 0
  Platelets Below (Month 7) | 0
  Red blood cells Above (Day 0) | 0
  Red blood cells Below (Day 0) | 1
  Red blood cells Above (Month 7) | 0
  Red blood cells Below (Month 7) | 0
  Total protein Above (Day 0) | 0
  Total protein Below (Day 0) | 8
  Total protein Above (Month 7) | 0
  Total protein Below (Month 7) | 3
  Total bilirubin Above (Day 0) | 2
  Total bilirubin Below (Day 0) | 0
  Total bilirubin Above (Month 7) | 4
  Total bilirubin Below (Month 7) | 0
  White blood cells Above (Day 0) | 0
  White blood cells Below (Day 0) | 1
  White blood cells Above (Month 7) | 0
  White blood cells Below (Month 7) | 5

ADVERSE EVENTS:
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 100/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=100)
Nasopharyngitis (Infections and infestations) | 18
Injection site pruritus (General disorders) | 16
Injection site warmth (General disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 6
Dysmenorrhoea (Reproductive system and breast disorders) | 6
Pain (General disorders) | 98
Redness (General disorders) | 85
Swelling (General disorders) | 81
Arthralgia (General disorders) | 15
Fatigue (General disorders) | 40
Fever (General disorders) | 10
Gastrointestinal symptoms (General disorders) | 17
Headache (General disorders) | 33
Myalgia (General disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.